CLINICAL TRIAL: NCT06469944
Title: A Phase 1/2 Open-Label, Umbrella Platform Design Study of Investigational Agents With Pembrolizumab (MK-3475) and Chemotherapy in Participants With 1L Locally Advanced Unresectable/Metastatic Gastroesophageal Adenocarcinoma (Gastric Adenocarcinoma, Gastroesophageal Junction Adenocarcinoma, and Esophageal Adenocarcinoma): Substudy 06C
Brief Title: Substudy 06C: A Study of Investigational Agents With Pembrolizumab (MK-3475) and Chemotherapy in Participants With First-Line Locally Advanced Unresectable/Metastatic Gastroesophageal Adenocarcinoma (MK-3475-06C/KEYMAKER-U06)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-06C; MK-3475-06C (Other: MSD); KEYMAKER-06C (Other: MSD); 2023-509307-33-00 (Registry Identifier: EU CT); U1111-1299-8084 (Registry Identifier: UTN)
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gastroesophageal Junction; Gastroesophageal Adenocarcinoma; Esophageal Neoplasms; Esophageal Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Capecitabine; Leucovorin; Levoleucovorin; Fluorouracil; Oxaliplatin; patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab plus Chemotherapy (Active Comparator): Participants will receive pembrolizumab 400 mg via intravenous (IV) injection on day 1 of every 6 week cycle (Q6W) for up to 18 cycles (up to ~2 years) AND investigator's choice of CAPOX chemotherapy (capecitabine 1000 mg/m^2 orally twice daily for 14 days every 3 weeks (Q3W) and oxaliplatin 130 mg/m^2 via IV infusion Q3W) OR mFOLFOX6 chemotherapy (oxaliplatin 85 mg/m^2 via IV infusion Q3W; 5-Fluorouracil (5-FU) 400 mg/^2 via bolus IV plus 2400 mg/m^2 continuous IV once every 2 weeks (Q2W); and leucovorin 400 mg/m^2 via IV infusion Q2W OR levoleucovorin 200 mg/m^2 Q2W).
  Interventions: Biological: Pembrolizumab; Drug: Capecitabine; Drug: Leucovorin; Drug: Levoleucovorin; Drug: 5-Fluorouracil (5-FU); Drug: Oxaliplatin
- Pembrolizumab plus Sacituzumab Tirumotecan plus Chemotherapy (Experimental): Participants will receive sacituzumab tirumotecan via IV infusion on Days 1, 15, and 29 Q6W until discontinuation, pembrolizumab 400 mg via IV injection on day 1 Q6W for up to 18 cycles (up to ~2 years) AND investigator's choice of capecitabine 1000 mg/m^2 orally twice daily for 14 days Q3W OR 5-FU 400 mg/^2 via bolus IV plus 2400 mg/m^2 continuous IV once Q2W AND leucovorin 400 mg/m^2 via IV infusion Q2W OR levoleucovorin 200 mg/m^2 Q2W.
  Interventions: Biological: Pembrolizumab; Biological: Sacituzumab Tirumotecan (sac-TMT); Drug: Capecitabine; Drug: Leucovorin; Drug: Levoleucovorin; Drug: 5-Fluorouracil (5-FU)
- Pembrolizumab plus Patritumab Deruxtecan plus Chemotherapy (Experimental): Participants will receive patritumab deruxtecan via IV infusion on Days 1 and 22 Q6W until discontinuation, pembrolizumab 400 mg via IV injection on day 1 Q6W for up to 18 cycles (up to ~2 years) AND investigator's choice of capecitabine 1000 mg/m^2 orally twice daily for 14 days Q3W OR 5-FU 400 mg/^2 via bolus IV plus 2400 mg/m^2 continuous IV once Q2W AND leucovorin 400 mg/m^2 via IV infusion Q2W OR levoleucovorin 200 mg/m^2 Q2W.
  Interventions: Biological: Pembrolizumab; Drug: Capecitabine; Drug: Leucovorin; Drug: Levoleucovorin; Drug: 5-Fluorouracil (5-FU); Biological: Patritumab Deruxtecan

INTERVENTIONS:
Biological: Pembrolizumab — Administered via intravenous (IV) infusion.
  Other Names: MK-3475; Keytruda®
Biological: Sacituzumab Tirumotecan (sac-TMT) — Administered via IV infusion.
  Other Names: MK-2870; SKB264
  Arms: Pembrolizumab plus Sacituzumab Tirumotecan plus Chemotherapy
Drug: Capecitabine — Administered via oral tablet.
  Other Names: XELODA
Drug: Leucovorin — Administered via IV infusion.
  Other Names: calcium folinate; folinic acid; WELLCOVORIN®
Drug: Levoleucovorin — Administered via IV infusion.
  Other Names: calcium levofolinate; levofolinic acid; FUSILEV®
Drug: 5-Fluorouracil (5-FU) — Administered via IV infusion
  Other Names: ADRUCIL®
Drug: Oxaliplatin — Administered via IV infusion
  Arms: Pembrolizumab plus Chemotherapy
Biological: Patritumab Deruxtecan — Administered via IV infusion
  Other Names: HER3-DXd; MK-1022; U3-1402
  Arms: Pembrolizumab plus Patritumab Deruxtecan plus Chemotherapy

SUMMARY:
This is a phase 1/2, multicenter, open-label umbrella platform study that will evaluate the safety and tolerability of investigational agents with pembrolizumab and fluoropyrimidine chemotherapy for the first-line (1L) treatment of participants with locally advanced unresectable or metastatic human epidermal growth factor receptor 2 (HER2)-negative gastric, gastroesophageal junction, or esophageal adenocarcinoma.

This substudy will have two phases: a safety lead-in phase and an efficacy phase. The safety lead-in phase will be used to evaluate the safety and tolerability, and to establish a recommended Phase 2 dose (RP2D) for investigational agents in combination with chemotherapy and immunotherapy. There is no formal hypothesis in this study.

DETAILED DESCRIPTION:
The master protocol is MK-3475-U06.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically and/or cytologically confirmed diagnosis of previously untreated locally advanced unresectable or metastatic first-line (1L) gastroesophageal adenocarcinoma
* Is not expected to require tumor resection during the treatment course
* Tumor tissue must be confirmed as negative for human epidermal growth factor receptor 2 (HER2) expression as classified by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines
* Core/excisional biopsy of a tumor lesion not previously irradiated has been provided
* Participants who have adverse events (AEs) due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline
* Participants with endocrine-related AEs who are adequately treated with hormone replacement therapy are eligible
* Has adequate organ function
* Has measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as determined by the local site investigator/radiology assessment and verified by blinded independent central review (BICR)
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 3 days prior to the first dose of study intervention
* Has a life expectancy of at least 6 months
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to allocation/randomization
* Participants with history of Hepatitis C Virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Human Immunodeficiency Virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has squamous cell or undifferentiated gastroesophageal cancer.
* Has had previous therapy for locally advanced unresectable or metastatic gastric/gastroesophageal junction (GEJ)/esophageal adenocarcinoma
* Has experienced weight loss >20% over 3 months before the first dose of study intervention
* Has a history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has Grade ≥2 peripheral neuropathy
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease within 6 months preceding study intervention
* Has accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to enrollment
* Has history of human immunodeficiency virus (HIV) infection with Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has received prior treatment with a trophoblast antigen 2 (TROP2)-targeted or anti-human epidermal growth factor receptor 3 (HER3) targeted agents
* Has received prior treatment with a topoisomerase I inhibitor-based antibody-drug conjugate (ADC) and/or a topoisomerase I inhibitor-based chemotherapy
* Has received prior systemic anticancer therapy within 4 weeks before the first dose of study intervention
* Has received prior therapy with an anti-Programmed Cell Death Protein 1 (PD-1), anti-Programmed Cell Death-Ligand 1 (PD-L1), anti-Programmed Cell Death-Ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (TCR)
* Has received prior radiotherapy within 2 weeks of start of study intervention, or has radiation related toxicities, requiring corticosteroids
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received a strong inducer/inhibitor of CYP3A4 that cannot be discontinued
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has Severe hypersensitivity (≥Grade 3) to pembrolizumab, sacituzumab tirumotecan, patritumab deruxtecan, or other biologic therapy, chemotherapy (ie, oxaliplatin, fluorouracil, capecitabine), leucovorin, levoleucovorin, or any of their excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has history of (noninfectious) pneumonitis or interstitial lung disease (ILD) that required steroids or has current pneumonitis or ILD, or where suspected ILD or pneumonitis cannot be ruled out by imaging at screening
* Has an active infection requiring systemic therapy
* Has concurrent active hepatitis B (defined as Hepatitis B surface antigen [HBsAg] positive and/or detectable HBV DNA) and hepatitis C virus (defined as anti-hepatitis C virus [HCV] Ab positive and detectable HCV ribonucleic acid [RNA] infection or a known history of hepatitis B and/or C infection
* Has history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's ability to cooperate with the requirements of the study
* Has gastrointestinal (GI) obstruction, poor oral intake, or difficulty in taking oral medication
* Has poorly controlled diarrhea
* Has had a major surgery or significant traumatic injury within 4 weeks before the first dose of study intervention
* Has history of allogeneic tissue/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2029-09-12 (Estimated); Study Completion 2029-09-12 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-in Phase: Number of Participants Who Experience One or More Dose-Limiting Toxicities (DLTs) | Up to approximately 28 days
  DLTs are defined as any drug-related adverse event (AE) according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) Version 5.0, observed during the DLT evaluation period that results in a change to a given dose or a delay in initiating the next cycle. The percentage of participants who experience at least one DLT will be reported.
Safety Lead-in Phase: Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 28 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Safety Lead-in Phase: Number of Participants Who Discontinued Study Intervention Due to an AE | Up to approximately 28 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 28 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) per RECIST 1.1 as Assessed by BICR | Up to approximately 55 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 55 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 55 months
  OS is defined as the time from randomization to the date of death from any cause.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 55 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 55 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Incidence of Antidrug Antibodies (ADA) to investigational agents - (sacituzumab tirumotecan (sac-TMT, MK-2870) and patritumab deruxtecan (HER3-DXd)) | At designated timepoints up to approximately 55 months
  Blood samples collected at designated timepoints will be used to determine the ADA response to investigational agents. The incidence of ADAs over time will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (42):
- United States (8):
  - University of Arizona Cancer Center-University of Arizona Cancer Center ( Site 6927), Tucson, Arizona
  - UCLA Hematology/Oncology - Santa Monica ( Site 6905), Los Angeles, California
  - Norton Hospital-Norton Cancer Institute - Downtown ( Site 6900), Louisville, Kentucky
  - The Cancer and Hematology Centers ( Site 6912), Grand Rapids, Michigan
  - Hematology-Oncology Associates of Central NY, P.C. ( Site 6925), East Syracuse, New York
  - Columbia University Irving Medical Center-CUIMC Herbert Irving Comprehensive Cancer Center Clinical ( Site 6907), New York, New York
  - UPMC Hillman Cancer Center-UPMC ( Site 6904), Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center ( Site 6920), Houston, Texas
- Brazil (3):
  - Liga Norte Riograndense Contra o Câncer ( Site 6303), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição ( Site 6301), Porto Alegre, Rio Grande do Sul
  - IBCC - Instituto Brasileiro de Controle do Câncer ( Site 6304), São Paulo
- Chile (7):
  - Clínica Puerto Montt ( Site 6409), Port Montt, Los Lagos Region
  - Centro de Investigación del Maule ( Site 6408), Talca, Maule Region
  - FALP-UIDO ( Site 6400), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión-Oncology ( Site 6404), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 6405), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 6401), Santiago, Region M. de Santiago
  - Bradford Hill Norte ( Site 6407), Antofagasta
- China (8):
  - Beijing Cancer hospital-Digestive Oncology ( Site 5500), Beijing, Beijing Municipality
  - The 900th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army ( Site 5501), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 5503), Xiamen, Fujian
  - Henan Cancer Hospital ( Site 5504), Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University ( Site 5514), Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center ( Site 5513), Shanghai, Shanghai Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi ( Site 5506), Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine ( Site 5510), Hangzhou, Zhejiang
- France (3):
  - CHU-BREST Cavale Blanche ( Site 5104), Brest, Finistere
  - CIC. ( Site 5100), Lille, Nord
  - Pitie Salpetriere University Hospital-Hepato-Gastro-Enterology ( Site 5102), Paris, Île-de-France Region
- Germany (2):
  - Universitaetsklinikum Duesseldorf-Gastroenterology, Hepatology and Infectiology ( Site 6802), Düsseldorf, North Rhine-Westphalia
  - Facharztzentrum Eppendorf-Facharztzentrum Eppendorf ( Site 6807), Hamburg
- Italy (2):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 5207), Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 5200), Milan, Lombardy
- Oslo universitetssykehus, Radiumhospitalet ( Site 6501), Oslo, Norway
- South Korea (2):
  - Asan Medical Center-Department of Oncology ( Site 5901), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 5900), Seoul
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 6701), Geneva, Canton of Geneva
  - Kantonsspital Graubünden-Medizin ( Site 6700), Chur, Kanton Graubünden
- Taiwan (4):
  - China Medical University Hospital ( Site 6007), Taichung
  - National Cheng Kung University Hospital ( Site 6001), Tainan
  - National Taiwan University Hospital-Oncology ( Site 6000), Taipei
  - Taipei Veterans General Hospital ( Site 6005), Taipei

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26339&tenant=MT_MSD_9011